CLINICAL TRIAL: NCT07324863
Title: The Effect of Ultrasound Guided External Oblique and Rectus Abdominis Plane Block (EXORA) on Neuroendocrine Stress Response in Adults Undergoing Umbilical Hernia Surgery: A Prospective Randomized Controlled Trial
Brief Title: Ultrasound Guided External Oblique and Rectus Abdominis Plane Block (EXORA) on Neuroendocrine Stress Response in Adults Undergoing Umbilical Hernia Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mayada Hady Mahmoud Sokeer, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD474/10/25
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Ultrasound; External Oblique; Rectus Abdominis Plane Block; Neuroendocrine Stress Response; Umbilical Hernia
MeSH Terms: conditions — Hernia, Umbilical | interventions — Anesthesia, General; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients will receive general anesthesia only.
  Interventions: Other: General anesthesia
- Group Ⅱ (Experimental): Patients will receive general anesthesia and an external oblique and rectus abdominis plane (EXORA) block with 0.25% bupivacaine.
  Interventions: Other: External oblique and rectus abdominis plane (EXORA) block

INTERVENTIONS:
Other: General anesthesia — Patients will receive general anesthesia only.
  Arms: Group I
Other: External oblique and rectus abdominis plane (EXORA) block — Patients will receive general anesthesia and an external oblique and rectus abdominis plane (EXORA) block with 0.25% bupivacaine.
  Arms: Group Ⅱ

SUMMARY:
This study aims to evaluate the efficacy of ultrasound-guided external oblique and rectus abdominis plane block on the neuroendocrine stress response and postoperative analgesia in adults undergoing umbilical hernia repair.

DETAILED DESCRIPTION:
Umbilical hernias of the abdomen are defined as a non-inguinal, non-hiatal defect in the fascia of the abdominal wall. Surgical stress response refers to the physiologic response to surgery and the hormonal and metabolic changes that follow it.

Fascial plane blocks are gaining attention for perioperative analgesia due to their efficacy and safety profiles. The external oblique and rectus abdominis plane (EXORA) block is an emerging technique that provides a sensory block to the anterolateral abdominal wall, potentially filling gaps left by other commonly used blocks, such as the quadratus lumborum (QLB) or erector spinae plane (ESP) blocks.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical status I and Ⅱ.
* Schedule for elective umbilical hernia surgery under general anesthesia.

Exclusion Criteria:

* ASA Ⅲ or Ⅳ.
* Patients with metabolic abnormalities, e.g., diabetes mellitus.
* Patients receiving corticosteroids.
* History of allergies to local anesthetics.
* Bleeding or coagulation disorders.
* Anatomical abnormalities.
* Psychiatric and neurological disorders.
* Complicated hernial defect (obstructed).
* Patient refusal.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Neuroendocrine stress response | 24 hours postoperatively
  Neuroendocrine stress response will be measured by blood glucose level in adults undergoing umbilical hernia repair.

SECONDARY OUTCOMES:
Serum cortisol level | 24 hours postoperatively
  Serum cortisol level will be measured.
Time of first rescue analgesia | 24 hours postoperatively
  Time of first rescue analgesia will be recorded from the end of surgery till first dose of morphine administration.
Total intraoperative fentanyl consumption | Intraoperatively
  Rescue dose of intraoperative fentanyl given will be recorded.
Total morphine consumption | 24 hours postoperatively
  Intravenous morphine (rescue analgesic) at a dosage of 3 mg will be administered when the Numerical Rating Scale (NRS) score will be ≥ 4. The total morphine consumption over a 24-hours period will be recorded for these individuals.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed in postoperative pain assessment using the Numerical Rating Scale (NRS), ranging from 0 to 10 (0 = "no pain," 10 = "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU),1,2,4,6,12,24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.